CLINICAL TRIAL: NCT05218759
Title: Exosomes Detection for the Prediction of the Efficacy and Adverse Reactions of Anlotinib in Patients With Advanced NSCLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: 3D Medicines (Industry)
Responsible Party: Principal Investigator, Aiqin Gu, Chief physician, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KS(Y)21217
Record Dates: First submitted 2022-01-19; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Anlotinib; Non-Small Cell Lung Cancer; exosome; detection biomarker
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm A (Experimental): Progressive disease (PD) after anlotinib administration
  Interventions: Drug: Anlotinib
- arm B (Experimental): Stable disease (SD) after anlotinib administration
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — anlotinib administration at a dose of 10 mg daily
  Other Names: H20180004

SUMMARY:
Exosomes detection for the prediction of the efficacy and adverse reactions of Anlotinib in patients with advanced NSCLC

DETAILED DESCRIPTION:
Explore blood exosomal miRNA as a biomarker for predicting the efficacy or risk of serious adverse reactions in patients with advanced lung adenocarcinoma (or lung squamous cell carcinoma) after anlotinib treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have signed informed consent.
2. Male or female, age between 18-75 years old.
3. Patients with advanced lung adenocarcinoma who failed standard treatment.
4. Complete prognostic assessment information.
5. Efficacy evaluation: PR/SD/PD.
6. Anlotinib single drug administration.
7. ECOG PS score: 0-1.
8. Patient's expected survival time is greater than 12 weeks.
9. The functions of main organs meets the following criteria: 1) absolute neutrophil count (ANC) ≥1.5×10^9/L; 2) white blood cell count (WBC) ≥3.0×10^9/L; 3) platelet (PLT) ≥100×10^9/L; 4) hemoglobin (Hb) ≥90g/L; 5); creatinine clearance ≥50ml/min or serum creatinine (Cr) ≤1.5×upper limit of normal (ULN); 6)serum total bilirubin (TBIL) ≤1.5×ULN; 7) alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN; 8) left ventricular ejection fraction (LVEF) ≥ the lower limit of the normal (50%); 9) Serum Cr ≤ 1.5ULN or creatinine clearance (CCr) ≥ 60ml / min; 10) ALT and AST ≤ 5ULN; 11) activated partial coagulation activity Enzyme time (APTT), international normalized ratio (INR), prothrombin time (PT)≤1.5×ULN.
10. Women of childbearing age should make sure their pregnancy test is negative within 2 weeks before the study, and keep using contraceptive methods during the study and within 24 weeks after the last administration of Anlotinib. For men, they must agree to use contraceptive methods during the study period and also 24 weeks after the last administration of Anlotinib.

Exclusion Criteria:

1. Patients whose plasma is not qualified for the test (hemolysis, precipitation, etc.)
2. Patients who have used Anlotinib before.
3. Pathological diagnosis results do not meet the requirements for entry.
4. Patients never used TKIs.
5. Patients with hemoptysis, more than 50mL per day.
6. Patients with other kinds of malignancies within 5 years.
7. Patients who have taken systemic therapy (immunotherapy, cytotoxic therapy, or other targeted therapies) within 6 weeks before grouping.
8. Patients who have symptoms of diseases that affect the patient's medication.
9. Patients who have suffered non-relieving toxicity from previous treatment.
10. Patients who have habitus of hemorrhage; the history of ulcer or fracture and non healing wounds.
11. Patients who have suffered arterial/venous thrombosis within 24 weeks.
12. Patients who have been diagnosed with mental disorder.
13. Patients who have suffered other diseases that may affect the patient's life safety and the results of this experiment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-21 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
PD | at the time of 2 months (2 cycles after treatment)
  Progressive disease (PD) after anlotinib administration
SD | at the time of 2 months (2 cycles after treatment)
  Stable disease (SD) after anlotinib administration

SECONDARY OUTCOMES:
Severe adverse reaction group | at the time of 2 months (2 cycles after treatment)
  Severe adverse reaction group after anlotinib administration
Adverse reaction non-serious group | at the time of 2 months (2 cycles after treatment)
  Adverse reaction non-serious group after anlotinib administration

CONTACTS AND LOCATIONS:
Overall Officials: Aiqin Gu, Chief physician, Principal Investigator — Shanghai Chest Hospital, Shanghai, China, 200030

IPD SHARING:
Plan to Share IPD: No